CLINICAL TRIAL: NCT05732038
Title: Using Mobile Technology to Reduce Stress in Caregivers of Persons With Dementia. A Scalable Solution to a Growing Problem.
Brief Title: STRIDE: Stress Reduction in Dementia Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ana-Maria Vranceanu, PhD, Associate Professor/Director, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022P001601
Record Dates: First submitted 2023-01-20; First posted 2023-02-16 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2024-01

CONDITIONS: Caregiver Stress
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy Minds Program (HMP) (Experimental): Participants assigned to the HMP group will be asked to practice 10 minutes per day for 12 weeks. The first four weeks will be prescribed. Weeks 5-12 will allow full access to the app's library.
  Interventions: Behavioral: Healthy Minds Program (HMP)
- Wellness App (WA) (Experimental): Participants in the WA group will be asked to listen to the app content for 10 minutes per day for the entire 12 weeks.
  Interventions: Behavioral: Wellness App (WA)

INTERVENTIONS:
Behavioral: Healthy Minds Program (HMP) — Participants assigned to the HMP group will be asked to complete a minimum of 10 minutes per day of meditation for 12 weeks. For the first four weeks, participants will listen to prescribed meditations that will teach them the foundations of mindfulness. During weeks 5-12, participants will have full access to the HMP meditation library.
  Arms: Healthy Minds Program (HMP)
Behavioral: Wellness App (WA) — Participants in the WA group will listen to a minimum of 10 minutes per day of a caregiver specific educational podcast (including topics such as "Caring for the Caregiver" or "Folate and Preventing Alzheimer's") delivered via a mobile app for the 12 weeks. The app contains one podcast per day for twelve weeks.
  Arms: Wellness App (WA)

SUMMARY:
The investigators aim to conduct a feasibility, proof of concept randomized controlled trial (RCT) of a smartphone app intervention (Healthy Minds Program; HMP) versus Wellness app (WA) among heterogeneous stressed caregivers of individuals with Alzheimer's disease and related dementias (ADRD). The investigators will test its feasibility (primary outcomes) and its preliminary effect in improvement in caregiver stress, emotional distress (depression and anxiety), and mindfulness. Participants will be randomized to one of the two conditions described above

DETAILED DESCRIPTION:
Using the NIA 2 year R21 grant mechanisms, we will examine the feasibility (markers of acceptability and demand), and proof of concept of Healthy Minds Program (HMP) versus Wellness App (WA) in decreasing stress and emotional distress in heterogeneous, geographically diverse, stressed caregivers of individuals with Alzheimer's disease and related dementias (ADRD). Participants in each arm will be asked to practice for 10 min/day.

To achieve our aims, we will conduct a single blind, pilot, feasibility, proof of concept randomized controlled trial (RCT) of HMP (12 weeks, > 10 minutes daily) versus WA; 12 weeks, >10 minutes daily). Assessments will be conducted at baseline, post program (12 weeks later) and at 20 weeks follow-up (~2 months after post-test). Caregivers will also complete weekly assessments.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. English fluency and literacy
3. Meeting criteria for being a caregiver (e.g., family or friend of a care recipient who provides unpaid care)
4. Perceived Stress Scale (4 items) version >= 6
5. Willing to be randomized
6. Care recipient must score >1 on the functional assessment scale (FAST)

Exclusion Criteria:

1. Any planned change in psychotropic pharmacologic treatment for the duration of the study
2. Use of any consumer-based mindfulness meditation app for more than 60 min/month in the past 6 months.
3. Current participation in a meditation program (e.g., mindfulness-based stress reduction, mindfulness-base cognitive therapy, etc.)
4. Major illness known to worsen dramatically or require surgery in the next 20 weeks (study duration)
5. Active treatment for cancer (chemotherapy, radiation)
6. Imminent placement of care recipient in a nursing home or with another caregiver (within 4 months).
7. Involvement in another clinical trial for caregivers.
8. For participants age 65 and older: four or more errors on the Short Portable Mental Status questionnaire (SPMSQ)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
Feasibility of Recruitment | 0 weeks
  We will assess number of dementia caregivers enrolled from the number of caregivers that were eligible. Our primary aim focuses on feasibility of recruitment during the trial.
Adherence to one of the two apps | 12 weeks
  We will assess data from the Healthy Minds Program app and the Podcast app to measure adherence to the intervention and the control conditions. Our benchmark will be that >=70% of caregivers will complete >=75% of weekly prescribed minutes (>=10 minutes/day).
Credibility and Expectancy Questionnaire (CEQ) | 0 weeks
  We will use the Credibility and Expectancy Questionnaire (CEQ) to assesses caregivers perceptions that the treatment will work after learning about the study. Scores range from 3-27; higher ratings indicate more belief that the program is logical and will help with the intended outcome.
Client Satisfaction Questionnaire (CSQ-3) | 12 weeks
  This will be used to assess caregivers' satisfaction with the intervention. Scores range from 3 to 12, with higher values indicating higher satisfaction.
Perceptions of daily meditations/podcast | 12 weeks
  We will assess caregivers' perception of their app's prescription by asking, "Do you think that the amount of daily prescribed app content was: too little, just enough, or too much?"
Perceptions of emails and text reminders | 12 weeks
  We will assess caregivers' perception of emails and text message reminders by asking, "Do you think that the amount of emails/texts you received was: too little, just enough, too much?"
Perceptions of the overall study | 12 weeks
  We will assess caregivers' perceptions of the study by asking, "Do you have any feedback about your experience in this program (content of the program, content of the text message reminders, etc.) that you would like to share?"
Feasibility of weekly Research Electronic Data Capture (RedCAP) measures | 12 weeks
  We will assess the feasibility of the weekly REDCap measures sent to patients by review of responses to ensure that >=70% caregivers will answer >=75%.
Perceptions of prompts/contacts in low adherence situations | 12 weeks
  We will assess caregivers' perception of the amount of prompts and contact in situations where they were not adhering to their practice by asking "Do you think that the amount of prompts you received when you struggled with your practice was: too little, just enough, too much?"
Feasibility of quantitative measures | 20 weeks
  We will assess the feasibility of the quantitative measures sent to caregivers with the benchmark of no questionnaires missing fully in >=25% caregivers.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | 0 weeks, 12 weeks, 20 weeks
  We will use the Hospital Anxiety and Depression Scale HADS, a 14-item measure that assesses symptoms of emotional distress (anxiety and depression). The anxiety and depression sub-scale are each scored from 0-21, with higher scores indicating greater severity of symptoms. Scores can be summed to create a global emotional distress score (0-42).
Applied Mindfulness Process Scale (AMPS) | 0 weeks, 12 weeks, 20 weeks
  We will use the Applied Mindfulness Process Scale (AMPS) to assess caregivers mindfulness. AMPS consists of 3 sub scales: de-centering, positive emotion regulation, and negative emotion regulation. Each sub scale is scored from 0-20. An overall score ranging from 0-60 can be obtained by summing all 15 items. Higher scores indicate greater mindfulness.
Stress Thermometer | 0-12 weeks, 20 weeks
  We will use a stress thermometer scale (0-10) to assess how caregivers rate their level of stress each week: "During the past week, how would you rate your stress on a scale from 0-10? (0 = not at all; 10 = extremely stressed)?"
Mindfulness Thermometer | 0-12 weeks, 20 weeks
  We will use a mindfulness thermometer scale (0-10) to assess how caregivers rate their level of mindfulness each week: "During the past week, how would you rate your mindfulness on a scale from 0-10? (0 = not at all; 10 = extremely mindful)?"
Emotional Distress Thermometer | 0-12 weeks, 20 weeks
  We will use an emotional distress thermometer scale (0-10) to assess how caregivers rate their level of distress each week: "During the past week, how would you rate your emotional distress on a scale from 0-10? (0 = not at all; 10 = extremely emotionally distressed)?"
Modified Patient Global Impression of Change (MPGI) | 12 weeks
  We will use the Modified Patient Global Impression of Change (MPGI), a 1-item questionnaire, to assess the extent to which caregivers perceive the intervention improved functioning and symptoms: "Do you think your ability to manage stress associated with caring for your loved one with dementia is now improved, about the same, or worse, as compared to before your participation in this program?"
Perceived Stress Scale 10 items (PSS-10) | 0 weeks, 12 weeks, 20 weeks
  We will use the PSS-10, to assess perceived stress using a 5-point Likert scale. Scores range from 0 to 40 with higher scores indicating greater stress.
Healthy Minds Index | 0 weeks, 12 weeks, 20 weeks
  This is a 17-item measure (each item is scored on a 0-4 scale) that assesses awareness (items 1-4; scored from 0-16), connection (items 5-10; scored from 0-24), insight (items 11-13; scored from 0-12), and purpose (items 14-17; scored from 0-16). Higher scores indicate greater levels of each sub scale.
Caregiver Reaction Scale | 0 weeks, 12 weeks, 20 weeks
  This measure assesses caregiver burden. We are administering the following sub scales: role entrapment (4 items); role overload (4 items); mastery as a caregiver (4 items); self mastery (4 items); workplace productivity (5 items). Each item is measured on 1-4 point scale. Sub scales with 4 items are scored from 4-16; sub scales with 5 items are scored from 5-20. Higher scores indicate higher levels of each sub scale's construct.

CONTACTS AND LOCATIONS:
Overall Officials: Ana-Maria Vranceanu, PhD, Principal Investigator — Massachusetts General Hospital; Jennifer Huberty, PhD, Principal Investigator — Mays Cancer Center at UT Health San Antonio MD Anderson
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Woodworth EC, Briskin EA, Plys E, Macklin E, Tatar RG, Huberty J, Vranceanu AM. Mindfulness-Based App to Reduce Stress in Caregivers of Persons With Alzheimer Disease and Related Dementias: Protocol for a Single-Blind Feasibility Proof-of-Concept Randomized Controlled Trial. JMIR Res Protoc. 2023 Oct 13;12:e50108. doi: 10.2196/50108. PMID 37831492